CLINICAL TRIAL: NCT05275452
Title: Assessing the Prevalence of Iodine Deficiency in Remote Communities of the Central Plateau, Haiti: a Cross-sectional Study (ARCH)
Brief Title: Prevalence of Iodine Deficiency in Remote Communities of Haiti
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Notre Dame (Other); Université Notre Dame d'Haiti UDERS de Hinche, Haiti (Unknown)
Responsible Party: Sponsor
Other Study IDs: ARCH
Record Dates: First submitted 2022-02-14; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Iodine Deficiency

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine samples will be retained for consenting participants for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- School age children aged 9-13 years
  Interventions: Other: No intervention
- Women of reproductive age aged 18-44 years
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Haiti is one of the few remaining countries that is at risk of iodine deficiency disorders. In the 2018 survey, iodized salt was found in <20% of households and iodine excretion from non-pregnant and pregnant women suggested inadequate intakes, with those in remote inland settings most at risk.

The Haiti Salt Program (HSP) was established in 2006 at the University of Notre Dame, US (UND). Using a self-sustaining business model that protects the livelihoods of all who work within it, the HSP has a goal of supplying fortified salt to combat IDD and lymphatic filariasis. HSP purchases salt from local small producers for processing in a local factory equipped with robust, standardized and controlled facilities that iodizes the salt under correct conditions, ready for fair resale to the consumer. The salt is currently distributed in the West Department, though a country-wide roll-out is envisaged. This initiative has the potential to accelerate optimization of population iodine intake across Haiti and through IDD prevention, positively contributing to the development of the country.

Data on iodine status and intake of native iodine-rich foods, iodized salt and other iodine-fortified foods e.g., bouillon cubes in Haiti, are sparse, particularly from rural and remote locations. An update on the situation in such remote areas in Haiti is trequired, to inform and leverage the development and implementation of iodized salt policy in the region.

The specific objective of this study is to assess the iodine status of two representative population subgroups, namely school-age children and women of reproductive age, in a remote region of the Central Plateau of Haiti. We hypothesize that the mUIC will indicate population iodine insufficiency in both of these population groups.

ELIGIBILITY:
We will recruit school age children (male and female, aged 9-13 years) and women of reproductive age (aged 18-44 years).

The inclusion criteria for all subjects will be:

1. residence within the study area for ≥12 months;
2. general good health as assessed by no reported treatment for chronic disease;
3. no known history of goiter or other thyroid disease;
4. no exposure to iodine containing contrast agent or medication within the last year;
5. Women of reproductive age should not currently be pregnant or be breastfeeding, assessed by asking the women.

Ages: 9 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The Central Plateau/Center Department is a predominantly rural Department in the Center/Northern part of Haiti. The Central Plateau is divided into the haut (upper) and bas (lower) plateau and covers an area of about 150 square miles (390 square km). The average elevation is about 1,000 feet (300 metres), and road access throughout the department is limited, with many areas accessible only by donkey/horse, motorcycle, or on foot. The Cahos Mountains form the western border of the department and the Noires Mountains form the southern border. Hinche is based largely on farming, raising of livestock, and trade.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Urinary iodine concentration | through study completion, estimated 2 to 3 months
  iodine measured in a spot sample of urine

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Rigutto, PhD, Principal Investigator — ETH Zürich
Locations (1):
- Université Notre Dame d'Haiti, Hinche, Haiti

IPD SHARING:
Plan to Share IPD: No